CLINICAL TRIAL: NCT04091139
Title: A Randomized-controlled Trial of a Locally Adapted Unified Protocol - Transdiagnostic Cognitive Behavioural Therapy for the Treatment of Common Mental Disorders in Adolescents in Hong Kong
Brief Title: Research of Unified Protocol for the Treatment of Common Mental Disorders in Adolescents in Hong Kong
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Castle Peak Hospital (Other Government)
Responsible Party: Principal Investigator, Sophie Yan Yan Cheung, Clinical Psychologist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPAHK01
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder; Anxiety Disorders
Keywords: Unified Protocol; Cognitive Behavioural Therapy; Depression; Anxiety; Adolescents
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is to examine the effect of transdiagnostic cognitive behavioural therapy (Unified Protocol for adolescents, UP-A), in comparison with treatment-as-usual, in the reduction of depressive and anxiety symptoms among adolescents with common mental disorders.
  All participants would be randomized into one of the two treatment arms, namely UP-A treatment condition (UP-A) and treatment-as-usual (TAU) condition. Following randomization, participants in UP-A condition would attend individual psychological treatment based on UP-A, which last for 10 to 12 weeks. Participants in the TAU condition would be provided with usual clinical psychological service (i.e. treatment as usual) in the first 12 weeks before they start attending the same individual treatment program based on UP-A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified protocol for adolescents (UP-A) (Experimental): The Unified Protocol (UP) is an emotion-focused, cognitive-behavioural intervention that is developed to target core temperamental characteristics underlying anxiety and depressive disorders. The goal of the UP is to help patients to cultivate a greater willingness to experience uncomfortable emotions and to reduce maladaptive emotion response tendencies, so as to lessen the intensity and frequency of uncomfortable emotions. Ehrenreich and colleagues modified from the original UP and developed the UP for adolescents (UP-A).
  A Chinese treatment protocol would be developed based on the UP-A. Contents of the treatment includes motivational enhancement, psychoeducation of emotion, avoidance and emotion driven behaviours, interoceptive exposure, cognitive reappraisal, emotion awareness training and emotion exposure. It consists of 10 to 12 individual sessions for the adolescents, and 4 to 6 sessions for parents or guardians.
  Interventions: Behavioral: Unified protocol for adolescents (UP-A)
- Treatment as usual (TAU) (Active Comparator): TAU participants will receive usual clinical psychological service provided in the clinic (i.e. treatment as usual) in the first 12 weeks, before they start receiving same individual treatment program based on UP-A.
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Unified protocol for adolescents (UP-A) — The Unified Protocol (UP) is an emotion-focused, cognitive-behavioural intervention that is developed to target core temperamental characteristics underlying anxiety and depressive disorders. The goal of the UP is to help patients to cultivate a greater willingness to experience uncomfortable emotions and to reduce maladaptive emotion response tendencies, so as to lessen the intensity and frequency of uncomfortable emotions. Ehrenreich and colleagues modified from the original UP and developed the UP for adolescents (UP-A).
  A Chinese treatment protocol would be developed based on the UP-A. Contents of the treatment includes motivational enhancement, psychoeducation of emotion, avoidance and emotion driven behaviours, interoceptive exposure, cognitive reappraisal, emotion awareness training and emotion exposure. It consists of 10 to 12 individual sessions for the adolescents, and 4 to 6 sessions for parents or guardians.
  Arms: Unified protocol for adolescents (UP-A)
Behavioral: Treatment as usual (TAU) — TAU participants will receive usual clinical psychological service provided in the clinic (i.e. treatment as usual) in the first 12 weeks, before they start receiving same individual treatment program based on UP-A.
  Arms: Treatment as usual (TAU)

SUMMARY:
The Unified Protocol (UP) is an emotion-focused, cognitive-behavioural intervention that is developed to target core temperamental characteristics underlying anxiety and depressive disorders. Ehrenreich and colleagues developed UP for adolescents (UP-A). The current study aims at evaluating efficacy of UP-A for the treatment of emotional disorders in Chinese adolescents in Hong Kong.

The current study would recruit 27 Chinese-speaking patients, age 13 to 18, with a primary diagnosis of any Diagnostic and Statistical Manual (Fifth edition) anxiety disorders and/or depressive disorder. They would be randomized into one of the two treatment arms, namely UP-A treatment condition (UP-A), and treatment-as-usual (TAU) condition. Following randomization, participants in the UP-A condition would attend individual treatment based on UP-A, which last for 10 to 12 weeks. Participants in the TAU condition would be provided with usual clinical psychological service (i.e. treatment as usual) in the first 12 weeks before they start attending the same individual treatment program.

Primary outcomes would be patient's self-rated measures on clinical symptoms, and secondary outcomes would be their clinical diagnoses, parent-rated and other self-rated measures. It is hypothesized that, comparing to those in TAU, participants in the UP-A condition would show improvements in depressive symptoms, anxiety symptoms and functional impairment at the end of treatment. When the outcomes of all participants are combined, it is hypothesized that participants will show demonstrate improvement in depressive symptoms, anxiety symptoms, and functional impairment after completing the UP-A and at the 3-month follow-up.

DETAILED DESCRIPTION:
A Chinese treatment protocol would be developed based on the UP-A. The adolescent program consists of 8 modules, and the parent program consists of 3 modules. Similar to the work by Ehrenreich and Barlow, a flexible modular approach would be adopted, when extra sessions would be arranged to cater for individual treatment needs and heterogeneity of symptom severity. The whole treatment comprised of 10 to 12 individual sessions for the adolescents, and 4 to 6 sessions for parents or guardian. The total duration would be around 3 months. Each treatment sessions would be around 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Age between 13 to 18 years.
* Primary diagnosis of any depression and/or anxiety disorders in fifth edition of the Diagnostic and Statistical Manual
* Use Chinese as primary written language
* For adolescents on medication, there must be 6-week stabilization period before study entry

Exclusion Criteria:

* Diagnoses of psychotic disorders, organic brain disease, bipolar disorder
* In high risk of self-harm or suicide
* Significant cognitive impairment (intellectual quotient lower than 80)
* Autism Spectrum Disorders
* Externalizing disorders with serious treatment interfering disruptive behavioural problems or substance abuse
* Attending concurrent psychotherapy
* Experience of attending a full-course of cognitive behavior therapy for anxiety or depression

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Change of depressive symptoms from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 12 (post-treatment) and Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 24 (post-treatment) and Week 36 (follow-up)
  Beck Depression Inventory for Youth (BDI-Y)
  * One of the inventories in the Beck Youth Inventories of Emotional and Social Impairment (Second Edition, Chinese version).
  * Construct measured: depressive symptoms.
  * Total scores would be converted into T-scores (range from 20-81) and descriptive classifications (normal, mild, moderate and severe) according to aged-norm.
  * The higher the T-scores, the more severe the depressive symptoms.
Change of anxiety symptoms from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 12 (post-treatment) and Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 24 (post-treatment) and Week 36 (follow-up)
  Beck Anxiety Inventory for Youth (BAI-Y)
  * One of the inventories in the Beck Youth Inventories of Emotional and Social Impairment (Second Edition, Chinese version).
  * Construct measured: anxiety symptoms.
  * Total scores would be converted into T-scores (range from 20-81) and descriptive classifications (normal, mild, moderate and severe) according to aged-norm.
  * The higher the T-scores, the more severe the anxiety symptoms.

SECONDARY OUTCOMES:
Change of psychiatric diagnosis of common mental disorders (based on fifth edition of Diagnostic and Statistical Manual) from baseline to treatment completion | UP-A: Week 0 (pre-treatment) and Week 12 (post-treatment); TAU: Week 0 (baseline), Week 12 (pre-treatment) and Week 24 (post-treatment)
  M.I.N.I. International Neuropsychiatric Interview for Children and Adolescent (MINIKID; English version 7.0.2)
  * Construct measured: psychiatric diagnoses.
  * Presence or absence of each of the following psychiatric diagnoses: major depressive disorder, bipolar disorder, panic disorder, agoraphobia, separation anxiety disorder, social anxiety disorder, specific phobia, obsessive-compulsive disorder, posttraumatic stress disorder, alcohol use disorder, substance use disorder, Tourette's disorder, attention-deficit/ hyperactivity disorder, conduct disorder, oppositional defiant disorder, psychotic disorder, anorexia nervosa, bulimia nervosa, binge eating disorder, generalized anxiety disorder, adjustment disorders and autism spectrum disorder.
Change of level of suicidality from baseline to treatment completion | UP-A: Week 0 (pre-treatment) and Week 12 (post-treatment); TAU: Week 0 (baseline), Week 12 (pre-treatment) and Week 24 (post-treatment)
  M.I.N.I. International Neuropsychiatric Interview for Children and Adolescent (MINIKID; English version 7.0.2) - Part B "Suicidality (for ages 13 through 17)"
  * Construct measured: suicidality.
  * Total scores (range from 0-169) which would be converted into descriptive classifications (low, moderate and high).
  * The higher the total scores, the higher the suicidality.
Change of functional impairment from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 12 (post-treatment) and Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 24 (post-treatment) and Week 36 (follow-up)
  Sheehan Disability Scale (SDS, 2012 version)
  * Construct measures: impairments in daily life.
  * Three separate impairment scores (each range from 0-10) on the domains of work/school, social life and family life/home responsibility.
  * The higher the impairment scores, the more the impairments.
Change of self-reported competencies and psychopathologies from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 12 (post-treatment) and Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 24 (post-treatment) and Week 36 (follow-up)
  Youth Self-report (YSR; 1991 & 2001 combined version, Chinese edition)
  * Construct measures: competencies and psychopathologies.
  * The competence scale consists of the activities and social subscales. Subscale total scores would be converted into T-scores (range from 20-55). A Total Competence Scale is computed from subscale scores, and would be converted into T-scores (range from 10-80). Descriptive classifications (normal, borderline and clinical) would be obtained from T-scores. The higher the T-score, the higher the competence.
  * The problem scale consists of the internalizing and externalizing problem subscales. Subscale total scores would be converted into T-scores (range from 26-100). A Total Problem Scale is computed from problem items, and would be converted into T-scores (range from 19-100). Descriptive classifications (normal, borderline and clinical) would be obtained from T-scores. The higher the T-score, the more severe the problems.
Change of parental-reported competencies and psychopathologies from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 12 (post-treatment) and Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 24 (post-treatment) and Week 36 (follow-up)
  Child Behavior Checklist (CBCL; 1991 & 2001 combined version, Chinese edition)
  * Construct measures: competencies and psychopathologies.
  * The competence scale consists of the activities, social and school subscales. Subscale total scores would be converted into T-scores (range from 20-55). A Total Competence Scale is computed from subscale scores, and would be converted into T-scores (range from 10-80). Descriptive classifications (normal, borderline and clinical) would be obtained from T-scores. The higher the T-score, the higher the competence.
  * The problem scale consists of the internalizing and externalizing problem subscales. Subscale total scores would be converted into T-scores (range from 29-100). A Total Problem Scale is computed from problem items, and would be converted into T-scores (range from 23-100). Descriptive classifications (normal, borderline and clinical) would be obtained from T-scores. The higher the T-score, the more severe the problems.
Change of depressive symptoms throughout the treatment, from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 1-12 (10-12 treatment sessions), Week 12 (post-treatment), Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 13-24 (10-12 treatment sessions), Week 24 (post-treatment), Week 36 (follow-up)
  Patient Health Questionnaire (PHQ-9)
  * Construct measured: depressive symptoms
  * Total scores (range from 0-27) and would be converted into descriptive classifications (normal, mild, moderate, moderately-severe and severe)
  * The higher the T-scores, the more severe the depressive symptoms
Change of anxiety symptoms throughout the treatment, from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 1-12 (10-12 treatment sessions), Week 12 (post-treatment), Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 13-24 (10-12 treatment sessions), Week 24 (post-treatment), Week 36 (follow-up)
  Generalized Anxiety Disorder Questionnaire (GAD-7)
  * Construct measured: anxiety symptoms
  * Total scores (range from 0-21) and would be converted into descriptive classifications (normal, mild, moderate, and severe)
  * The higher the T-scores, the more severe the anxiety symptoms
Change of self-reported problem severity throughout the treatment, from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 1-12 (10-12 treatment sessions), Week 12 (post-treatment), Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 13-24 (10-12 treatment sessions), Week 24 (post-treatment), Week 36 (follow-up)
  Subjective rating of distress (SUDS)
  * Construct measured: subjective rating of problem severity
  * Participants are asked to list up to a maximum of 3 problems, and give a subjective rating of distress for each of the problem listed. An average score (range from 0-10) would be calculated.
  * The higher the average score, the more severe the problems.
Change of parental-reported problem severity throughout the treatment, from baseline to treatment completion and at the three-month follow-up | UP-A: Week 0 (pre-treatment), Week 1-12 (4-6 parent sessions), Week 12 (post-treatment), Week 24 (follow-up); TAU: Week 0 (baseline), Week 12 (pre-treatment), Week 13-24 (4-6 parent sessions), Week 24 (post-treatment), Week 36 (follow-up)
  Subjective rating of distress - parents (SUDS - parents)
  * Construct measured: parental rating of problem severity
  * Parents are asked to list up to a maximum of 3 problems faced by the participants, and give a subjective rating of distress for each of the problem listed. An average score (range from 0-10) would be calculated.
  * The higher the average score, the more severe the problems.

OTHER OUTCOMES:
Self-reported subjective satisfaction towards treatment | UP-A: Week 12 (post-treatment); TAU: Week 24 (post-treatment)
  Satisfaction survey
  * Construct measured: subjective rating of satisfaction towards treatment
  * Participants are asked to give subjective ratings of how easy it is to apply the skills introduced in the treatment, and how useful these skills (range from 0-10). The higher the scores, the easier or more useful the application of skills respectively.
  * Participants would also complete discrete ratings of whether or not they are satisfied with the treatment duration and treatment intensity respectively, and whether or not they would recommend the program to others.
Parental-reported subjective satisfaction towards treatment | UP-A: Week 12 (post-treatment); TAU: Week 24 (post-treatment)
  Satisfaction survey (parents)
  * Construct measured: subjective rating of satisfaction towards treatment
  * Parents are asked to give subjective ratings of satisfaction of treatment. An average score (range from 0-10) would be calculated from these ratings. The higher the average score, the higher the level of satisfaction.
  * Parents would also complete discrete ratings of whether or not they are satisfied with the treatment duration and treatment intensity respectively, and whether or not they would recommend the program to others.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Yan Yan Cheung, MSocSc, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Psychology, The Chinese University of Hong Kong, Hong Kong, HK, Hong Kong

IPD SHARING:
Plan to Share IPD: No